CLINICAL TRIAL: NCT01664494
Title: A Non-Interventional Trial of Xeloda in Metastatic Colorectal Cancer, Adjuvant Colon Cancer, Advanced Gastric Cancer and Breast Cancer
Brief Title: An Observational Study of Xeloda (Capecitabine) in Patients With Metastatic Colorectal Cancer, Colon Cancer in the Adjuvant Setting, Advanced Gastric Cancer or Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25281
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer, Colorectal Cancer, Gastric Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Stomach Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Capecitabine: Participants will receive capecitabine according to the label text as monotherapy (1250 mg/m^2 twice daily) or combination therapy (800 to 1000 mg/m^2 or 1250 mg/m^2 twice daily) for 14 consecutive days followed by a treatment break of 7 days.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be given according to the label text as monotherapy (1250 mg/m^2 twice daily) or combination therapy (800 to 1000 mg/m^2 or 1250 mg/m^2 twice daily) for 14 consecutive days followed by a treatment break of 7 days.

SUMMARY:
This multi-center observational study will evaluate the use of Xeloda (capecitabine) in patients with metastatic colorectal cancer, colon cancer in the adjuvant setting, advanced gastric cancer and breast cancer in routine clinical practice. Eligible patients receiving treatment with Xeloda according to product label will be followed for up to 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic colorectal cancer, colon cancer in the adjuvant setting, advanced gastric cancer or breast cancer who are candidates for receiving Xeloda according to product label

Exclusion Criteria:

* Contraindications according to label and off-label use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients metastatic colorectal cancer, colon cancer in the adjuvant setting, advanced gastric cancer or breast cancer receiving Xeloda
Sampling Method: Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 563 participants were included from April 2010 to July 2012 at 21 sites in Austria.
Pre-assignment Details: Of 563 participants, 220 were treated for adjuvant colon cancer, 200 were treated for metastatic colorectal cancer, 84 were treated for metastatic breast cancer, and 59 were treated for advanced gastric cancer.
Groups:
- Capecitabine: Participants received capecitabine according to the label text as monotherapy (1250 mg/m^2 twice daily) or combination therapy (800 to 1000 mg/m^2 or 1250 mg/m^2 twice daily) for 14 consecutive days followed by a treatment break of 7 days.
Period: Overall Study
Arm/Group | Capecitabine
Started | 563
Completed | 370
Not Completed | 193
Not completed — Withdrawal by Subject | 27
Not completed — Death | 18
Not completed — Other | 49
Not completed — Lost to Follow-up | 99

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine
Number analyzed (Participants) | 563
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — The gender was not assessed in this study.
  Male | NA — The gender was not assessed in this study.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Routine Clinical Use of Capecitabine as Per the Line of Treatment
Description: Choice of line of treatment in adjuvant and advanced or metastatic cancer for capecitabine was observed.
Time Frame: Approximately 3 years; or up to disease progression, death or stop of capecitabine treatment, whichever occurred first
Population: All enrolled participants were considered for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 563
Participants
  Adjuvant therapy | 220
  First line therapy | 176
  Second line therapy | 89
  Third line therapy | 78

2. Secondary Outcome: Median Dose of Capecitabine
Description: Median dose of capecitabine for treatment of metastatic colorectal cancer, adjuvant colon cancer, advanced gastric cancer, or metastatic breast cancer in this study was presented.
Time Frame: Approximately 3 years; or up to disease progression, death or stop of capecitabine treatment, whichever occurred first
Population: All enrolled participants were considered for this outcome measure.
Measure: Median (Full Range); unit: Milligrams
Arm/Group | Capecitabine
Number analyzed (Participants) | 563
Milligrams
  Month 7 | 3500 [1500 to 5000]
  From Month 8 onwards | 3000 [900 to 5000]

ADVERSE EVENTS:
Time Frame: Approximately 3 years; or up to disease progression, death or stop of capecitabine treatment, whichever occurred first
Description: SAEs and other AEs were collected in all enrolled participants.
Arm/Group | Capecitabine
Serious Adverse Events (participants affected / at risk) | 34/563
Other Adverse Events (participants affected / at risk) | 271/563
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=563)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 7
Diverticulum intestinal (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 7
General physical health deterioration (General disorders) | 7
Multiple Organ Failure (General disorders) | 1
Sepsis (Infections and infestations) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Inflammatory marker increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypertonia (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5
Blister (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=563)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 172
Diarrhoea (Gastrointestinal disorders) | 117
Nausea (Gastrointestinal disorders) | 110
Stomatitis (Gastrointestinal disorders) | 63
Vomiting (Gastrointestinal disorders) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.